CLINICAL TRIAL: NCT05122546
Title: Pilot Study to Evaluate the Biologic Effect of CBM588 in Combination With Cabozantinib/Nivolumab for Patients With Metastatic Renal Cell Carcinoma
Brief Title: CBM588 in Combination With Nivolumab and Cabozantinib for the Treatment of Advanced or Metastatic Kidney Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21133; NCI-2021-05559 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21133 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2021-10-27; First posted 2021-11-16 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Advanced Clear Cell Renal Cell Carcinoma; Advanced Papillary Renal Cell Carcinoma; Advanced Renal Cell Carcinoma; Advanced Sarcomatoid Renal Cell Carcinoma; Metastatic Clear Cell Renal Cell Carcinoma; Metastatic Papillary Renal Cell Carcinoma; Metastatic Renal Cell Carcinoma; Metastatic Sarcomatoid Renal Cell Carcinoma; Stage III Renal Cell Cancer AJCC v8; Stage IV Renal Cell Cancer AJCC v8; Unresectable Clear Cell Renal Cell Carcinoma; Unresectable Renal Cell Carcinoma
MeSH Terms: conditions — Clear-cell metastatic renal cell carcinoma; Carcinoma, Renal Cell | interventions — cabozantinib; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 2 (CBM588, nivolumab, cabozantinib S-malate) (Experimental): Patients receive CBM588 PO BID, nivolumab IV over 30 minutes on day 1, and cabozantinib S-malate PO QD. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cabozantinib S-malate; Drug: Clostridium butyricum CBM 588 Probiotic Strain; Biological: Nivolumab
- Arm I (nivolumab, cabozantinib S-malate) (Active Comparator): Patients receive nivolumab IV over 30 minutes on day 1 and cabozantinib S-malate PO QD. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cabozantinib S-malate; Biological: Nivolumab

INTERVENTIONS:
Drug: Cabozantinib S-malate — Given PO
  Other Names: BMS-907351; Cabometyx; Cometriq; XL-184; XL184
Drug: Clostridium butyricum CBM 588 Probiotic Strain — Given PO
  Other Names: C. butyricum CBM 588 Probiotic Strain; C. butyricum MIYAIRI Strain; C. butyricum Strain MIYAIRI 588; CBM 588; CBM588; Clostridium butyricum MIYAIRI 588; Clostridium butyricum MIYAIRI 588 Probiotic Strain; MIYAIRI 588; MIYAIRI 588 Strain of C. butyricum
  Arms: Arm 2 (CBM588, nivolumab, cabozantinib S-malate)
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; CMAB819; MDX-1106; NIVO; Nivolumab Biosimilar CMAB819; ONO-4538; Opdivo

SUMMARY:
This phase I trial evaluates the effects of CBM588 in combination with standard therapies, nivolumab and cabozantinib, in treating patients with kidney cancer that has spread to other places in the body (advanced/metastatic). The digestive microbiome may have an effect on how patients respond to treatment, and previous research shows that a specific bacteria found in the gut (Bifidobacterium) may predispose participants to a better response to standard therapies. CBM588 is a strain of bacteria that can restore species of Bifidobacterium to the microbiome. The primary aim of this study is to determine how CBM588 changes the microbiome of patients with metastatic renal cell carcinoma. Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. cabozantinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving CBM588, nivolumab, and cabozantinib may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the effect of clostridium butyricum CBM 588 probiotic strain (CBM588) (in combination with cabozantinib/nivolumab) in modulation of the gut microbiome in patients with metastatic renal cell carcinoma (mRCC).

SECONDARY OBJECTIVES:

I. To evaluate the effect of CBM588 on the clinical efficacy of the cabozantinib/nivolumab combination.

II. To assess the effect of CBM588 on systemic immunodulation of the cabozantinib/nivolumab combination in patients with mRCC.

III. To assess the effect of CBM588 on toxicities such as diarrhea and nausea using Common Terminology Criteria for Adverse Events (CTCAE) version (v)5 criteria with the cabozantinib/nivolumab combination in patients with mRCC.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM 1: Patients receive nivolumab intravenously (IV) over 30 minutes on day 1 and cabozantinib S-malate orally (PO) once daily (QD). Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM 2: Patients receive CBM588 PO twice a day (BID), nivolumab IV over 30 minutes on day 1, and cabozantinib S-malate PO QD. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of renal cell carcinoma (RCC) with a clear-cell, papillary or sarcomatoid component
* Advanced (not amenable to curative surgery or radiation therapy) or metastatic (American Joint Committee on Cancer [AJCC] stage IV) RCC
* No prior systemic therapy for RCC with the following exception:

  * One prior adjuvant or neoadjuvant therapy for completely resectable RCC if recurrence occurred at least 6 months after the last dose of adjuvant or neoadjuvant therapy
* Measurable disease as per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Recovery to baseline or =< grade 1 CTCAE v5 from toxicities related to any prior treatments unless adverse events (AE[s]) are clinically nonsignificant and/or stable on supportive therapy
* Karnofsky performance status >= 70%
* Males and females, ages >= 18
* Any ethnicity or race
* Absolute neutrophil count (ANC) >= 1500/uL without granulocyte colony-stimulating factor support (within 14 days before first dose of study treatment)
* White blood cell count >= 2500/uL (within 14 days before first dose of study treatment)
* Platelets >= 100,000/uL without transfusion (within 14 days before first dose of study treatment)
* Hemoglobin >= 9 g/dL (>= 90 g/L) (within 14 days before first dose of study treatment)
* Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase (ALP) =< 3 x upper limit of normal (ULN). ALP =< 5 x ULN with documented bone metastases (within 14 days before first dose of study treatment)
* Total bilirubin =< 1.5 x ULN (for subjects with Gilbert's disease =< 3 x ULN) (within 14 days before first dose of study treatment)
* Serum albumin >= 2.8 g/dl (within 14 days before first dose of study treatment)
* Prothrombin time (PT)/international normalized ratio (INR) or partial thromboplastin time (PTT) test < 1.3 x the laboratory ULN (within 14 days before first dose of study treatment)
* Serum creatinine =< 1.5 x ULN or calculated creatinine clearance >= 40mL/min (>= 0.675 mL/sec) using the Cockcroft-Gault equation (within 14 days before first dose of study treatment)
* Urine protein/creatinine ratio (UPCR) =< 1 mg/mg (=< 113.2 mg/mmol), or 24-hour (h) urine protein =< 1 g (within 14 days before first dose of study treatment)
* Capable of understanding and complying with the protocol requirements and must have signed the informed consent document
* Sexually active fertile subjects and their partners must agree to use medically accepted methods of contraception (e.g., barrier methods, including male condom, female condom, or diaphragm with spermicidal gel) during the course of the study and for 4 months after the last dose of cabozantinib, 5 months after the last dose of nivolumab for women with childbearing potential, and 7 months after the last dose of nivolumab for men
* Female subjects of childbearing potential must not be pregnant at screening. Female subjects are considered to be of childbearing potential unless one of the following criteria is met: documented permanent sterilization (hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) or documented postmenopausal status (defined as 12 months of amenorrhea in a woman > 45 years-of-age in the absence of other biological or physiological causes. In addition, females < 55 years-of-age must have a serum follicle stimulating [FSH] level > 40 mIU/mL to confirm menopause). Note: Documentation may include review of medical records, medical examinations, or medical history interview by study site

Exclusion Criteria:

* Prior treatment with cabozantinib
* Current use, or intent to use, probiotics, yogurt, or bacterial fortified foods during the period of treatment
* Active interstitial lung disease (ILD)/pneumonitis or history of ILD/pneumonitis requiring treatment with systemic steroids
* Known medical condition (e.g., a condition associated with diarrhea or acute diverticulitis) that, in the investigator's opinion, would increase the risk associated with study participation or study drug administration or interfere with the interpretation of safety results
* Receipt of any type of small molecule kinase inhibitor (including investigational kinase inhibitor) within 2 weeks before first dose of study treatment
* Receipt of any type of cytotoxic, biologic, or other systemic anticancer therapy (including investigational) within 4 weeks before first dose of study treatment
* Radiation therapy for bone metastasis within 2 weeks or any other radiation therapy within 4 weeks before first dose of study treatment. Systemic treatment with radionuclides within 6 weeks before first dose of study treatment. Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible
* Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 4 weeks prior to first dose of study treatment after radiotherapy or at least 4 weeks prior to first dose of study treatment after major surgery (e.g., removal or biopsy of brain metastasis). Subjects must have complete wound healing from major surgery or minor surgery before first dose of study treatment. Eligible subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of first dose of study treatment
* Concomitant anticoagulation with coumarin agents (e.g., warfarin), direct thrombin inhibitors (e.g., dabigatran), direct factor Xa inhibitor betrixaban, or platelet inhibitors (e.g., clopidogrel). Allowed anticoagulants are the following:

  * Prophylactic use of low-dose aspirin for cardio-protection (per local applicable guidelines) and low-dose low molecular weight heparins (LMWH)
  * Therapeutic doses of LMWH or anticoagulation with direct factor Xa inhibitors rivaroxaban, edoxaban, or apixaban in subjects without known brain metastases who are on a stable dose of the anticoagulant for at least 1 week before first dose of study treatment without clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor
* Administration of a live, attenuated vaccine within 30 days before first dose of study treatment
* The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  * Cardiovascular disorders:

    * Congestive heart failure New York Heart Association class 3 or 4, unstable angina pectoris, serious cardiac arrhythmias
    * Uncontrolled hypertension defined as sustained blood pressure (BP) > 140 mm Hg systolic or > 90 mm Hg diastolic despite optimal antihypertensive treatment
    * Stroke (including transient ischemic attack [TIA]), myocardial infarction (MI), or other ischemic event, or thromboembolic event (e.g., deep venous thrombosis, pulmonary embolism) within 6 months before first dose of study treatment

      * Subjects with a diagnosis of incidental, subsegmental pulmonary embolism (PE) or deep vein thrombosis (DVT) within 6 months are allowed if stable, asymptomatic, and treated with a stable dose of permitted anticoagulation for at least 1 week before first dose of study treatment
  * Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation:

    * The subject has evidence of tumor invading the GI tract, active peptic ulcer disease, inflammatory bowel disease (e.g., Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis, acute obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction.
    * Abdominal fistula, GI perforation, bowel obstruction, or intra-abdominal abscess within 6 months before first dose of study treatment. Note: Complete healing of an intra-abdominal abscess must be confirmed before first dose of study treatment
* Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or other history of significant bleeding (e.g., pulmonary hemorrhage) within 12 weeks before first dose of study treatment
* Cavitating pulmonary lesion(s) or known endotracheal or endobronchial disease manifestation
* Lesions invading or encasing any major blood vessels
* Other clinically significant disorders that would preclude safe study participation:

  * Any active, known, or suspected autoimmune disease will be excluded, with the following exceptions:

    * Type 1 diabetes mellitus.
    * Hypothyroidism only requiring hormone replacement.
    * Skin disorders (e.g., vitiligo, psoriasis, or alopecia) not requiring systemic treatment.
    * Conditions not expected to recur in the absence of an external trigger.
  * Any condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days before first dose of study treatment.

    * Note: Inhaled, intranasal, intra-articular, or topical steroids are permitted. Adrenal replacement steroid doses > 10 mg daily prednisone equivalent are permitted. Transient short-term use of systemic corticosteroids for allergic conditions (e.g., contrast allergy) is also allowed.
  * Active infection requiring systemic treatment. Acute or chronic hepatitis B or C infection, known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness, or known positive test for tuberculosis infection where there is clinical or radiographic evidence of active mycobacterial infection.
  * History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan.
  * Serious non-healing wound/ulcer/bone fracture.
  * Malabsorption syndrome.
  * Uncompensated/symptomatic hypothyroidism.
  * Moderate to severe hepatic impairment (Child-Pugh B or C).
  * Requirement for hemodialysis or peritoneal dialysis.
  * History of solid organ or allogenic stem cell transplant.
* Major surgery (e.g., laparoscopic nephrectomy, GI surgery, removal, or biopsy of brain metastasis) within 2 weeks before first dose of study treatment. Minor surgeries within 10 days before first dose of study treatment. Subjects must have complete wound healing from major surgery or minor surgery before first dose of study treatment. Subjects with clinically relevant ongoing complications from prior surgery are not eligible.
* Corrected QT interval calculated by the Fridericia formula (QTcF) > 500 ms per electrocardiogram (ECG) within 14 days before first dose of study treatment. Furthermore, subjects with a history of additional risk factors for torsades de pointes (e.g., long QT syndrome) are also excluded.

  * Note: If a single ECG shows a QTcF with an absolute value > 500 ms, two additional ECGs at intervals of approximately 3 min must be performed within 30 min after the initial ECG, and the average of these three consecutive results for QTcF will be used to determine eligibility.
* Pregnant or lactating females
* Inability to swallow tablets or unwillingness or inability to receive IV administration
* Previously identified allergy or hypersensitivity to components of the study treatment formulations or history of severe infusion-related reactions to monoclonal antibodies. Subjects with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption are also excluded.
* Any other active malignancy at time of first dose of study treatment or diagnosis of another malignancy within 3 years prior to first dose of study treatment that requires active treatment, except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2026-01-27 (Estimated); Study Completion 2026-01-27 (Estimated)

PRIMARY OUTCOMES:
Change in Bifidobacterium composition of stool | Baseline to week 12 of therapy
  Will be assessed for patients' stool sample

SECONDARY OUTCOMES:
Comparison of the Shannon index (a measure of microbial diversity) | Baseline to week 12 of therapy
  Using translational methods, will compute the Shannon index at baseline for a comparison of microbial diversity.
Best overall response | Up to 2 years
  Will be assessed by Response Evaluation Criteria in Solid Tumors (RECIST) criteria. The association between treatment arm and overall response as per RECIST criteria (response observed versus not observed) will be examined using Fisher's exact test.
Progression-free survival | From enrollment to progression, assessed up to 2 years
  The difference in progression free survival across the two groups will be explored graphically using Kaplan-Meier survival plots. Median progression-free survival time for each of the two arms will be reported and Cox Proportional Hazards model will be used to estimate the hazard ratio and its confidence interval.
Proportion of circulating regulatory T-cells | Baseline up to 2 years
  Using translational methods will estimate the proportion of T-cells in the blood. This will be assessed graphically across serial timepoints of blood collection to ascertain any trends. Will compare the proportion of circulating T-cells with cabozantinib/nivolumab alone versus cabozantinib/nivolumab with CBM 588.
Change in proportion of circulating myeloid-derived suppressor cells (MDSC) | Baseline up to 2 years
  Using translational methods will estimate the proportion of MDSCs in the blood. This will be assessed graphically across serial timepoints of blood collection to ascertain any trends. Will compare the proportion of circulating MDSCs with cabozantinib/nivolumab alone versus cabozantinib/nivolumab with CBM 588.
Comparison of IL-6, IL-8 and other cytokines/chemokines | Baseline up to 2 years
  Using translational methods will estimate the proportion of serum cytokines in the blood. This will be assessed graphically across serial time points of blood collection to ascertain any trends. Will compare the IL-6, IL-8, and other cytokines/chemokines with cabozantinib/nivolumab alone versus cabozantinib/nivolumab with CBM 588.
Incidence of adverse events | Baseline up to 2 years
  Will compare toxicities, such as diarrhea and nausea, using Common Terminology Criteria for Adverse Events version 5 with cabozantinib/nivolumab alone versus cabozantinib/nivolumab with CBM 588.

CONTACTS AND LOCATIONS:
Overall Officials: Sumanta K Pal, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

REFERENCES:
- [Derived] Ebrahimi H, Dizman N, Meza L, Malhotra J, Li X, Dorff T, Frankel P, Llamas-Quitiquit M, Hsu J, Zengin ZB, Alcantara M, Castro D, Mercier B, Chawla N, Chehrazi-Raffle A, Barragan-Carrillo R, Jaime-Casas S, Govindarajan A, Gillece J, Trent J, Lee PP, Parks TP, Takahashi M, Hayashi A, Kortylewski M, Caporaso JG, Lee K, Tripathi A, Pal SK. Cabozantinib and nivolumab with or without live bacterial supplementation in metastatic renal cell carcinoma: a randomized phase 1 trial. Nat Med. 2024 Sep;30(9):2576-2585. doi: 10.1038/s41591-024-03086-4. Epub 2024 Jun 28. PMID 38942995